CLINICAL TRIAL: NCT07022314
Title: FIZE kUO® Real-Time Measurement of Urine Output Response to Fluid Therapy and Diuretics in Cardiovascular Surgery Patients: A Prospective Post-Market Study
Brief Title: Urine Output Response to Fluid and Diuretic Therapy in Cardiac ICU Patients Monitored With FIZE kUO®
Status: Not yet recruiting | Type: Observational
Sponsor: FIZE Medical ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: FM-01
Record Dates: First submitted 2025-06-04; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: AKI - Acute Kidney Injury; Cardiac Surgery; Fluid Therapy; Hemodynamic Instability; Postoperative Complications
Keywords: FIZE kUO; Urine Output; Fluid Management; Diuretics; Cardiothoracic Surgery
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cardiothoracic ICU Patients: Adult patients (≥18 years old) undergoing coronary artery bypass graft (CABG) and/or valve surgery, admitted postoperatively to the Cardiothoracic Intensive Care Unit (CTICU), and connected to the FIZE kUO® device for real-time urine output monitoring as part of standard care.
  Interventions: Device: FIZE kUO®

INTERVENTIONS:
Device: FIZE kUO® — FIZE kUO® is a commercially available, non-invasive device used for continuous, minute-by-minute real-time urine output monitoring in patients with an indwelling Foley catheter. In this observational study, the device is used during and after cardiac surgery as part of routine clinical care. Urine output data, along with additional clinical parameters, are collected throughout the study for research analysis.

SUMMARY:
This prospective observational study evaluates the real-time urine output response to fluid therapy and diuretics in cardiothoracic intensive care unit (CTICU) patients monitored with the FIZE kUO® device. The study aims to assess how continuous urine output monitoring can inform fluid management and improve patient outcomes post-cardiac surgery.

DETAILED DESCRIPTION:
The study involves adult patients undergoing coronary artery bypass graft (CABG) or valve replacement/repair surgeries. Utilizing the FIZE kUO® device, continuous urine output data will be collected to analyze responses to hemodynamic interventions, including fluid boluses and diuretics. Secondary objectives include assessing urine output differences in patients with and without postoperative acute kidney injury (AKI), responses to vasopressors, and capturing real-time urine output data from FIZE kUO® for observational analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older scheduled for CABG or valve surgery and expected postoperative admission to CTICU
2. Ability to provide informed consent

Exclusion Criteria:

1. Pregnancy
2. Preoperative dialysis (chronic or acute)
3. Enrollment in other interventional trials assessing urine output or AKI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients in the cardiothoracic ICU who require continuous urine output monitoring and are connected to the FIZE kUO® device as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Urine output response to fluid boluses and diuretics | 4 hours (2 hours before and 2 hours after intervention)
  Change in urine output measured by FIZE kUO® during 2 hours before and after fluid or diuretic administration.

SECONDARY OUTCOMES:
Difference in urine output during surgery between patients with and without AKI | Perioperative/Periprocedural
  Comparison of urine output measured by FIZE kUO® in patients who develop AKI vs. those who do not
Urine output response to vasopressors | 4 hours (2 hours before and 2 hours after intervention)
  Change in urine output measured by FIZE kUO® before and after vasopressor administration
Evaluation of FIZE kUO® Urine Output Monitoring Compared to Manual Measurement | Through ICU stay, up to 5 days
  Comparison of FIZE kUO® urine output with manual measurement of urine output

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel